CLINICAL TRIAL: NCT05310253
Title: "Fight-or-flight" Versus "tend-and-befriend" Response to Behavioral and Pharmacological Interventions in Patients with Borderline Personality Disorder (Part II)
Brief Title: Stress & Social Cognition in BPD (part 2)
Acronym: SOKO-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Katja Wingenfeld, "Fight-or-flight" versus "tend-and-befriend" response to behavioral and pharmacological interventions in patients with borderline personality disorder, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: WI 3396/12-1.2
Record Dates: First submitted 2022-03-14; First posted 2022-04-04 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Fludrocortisone; Psychological Tests

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Fludrocortisone & TSST - BPD patients (Experimental): intake of 0.4mg fludrocortisone (orally) before stress
  Interventions: Drug: Fludrocortisone; Behavioral: Trier Social Stress Test (TSST)
- Fludrocortisone & TSST - Healthy controls (Experimental): intake of 0.4mg fludrocortisone (orally) before stress
  Interventions: Drug: Fludrocortisone; Behavioral: Trier Social Stress Test (TSST)
- Placebo pills & TSST - BPD patients (Experimental): intake of placebo pill before stress
  Interventions: Drug: Placebo; Behavioral: Trier Social Stress Test (TSST)
- Placebo pills & TSST - Healthy controls (Experimental): intake of placebo pill before stress
  Interventions: Drug: Placebo; Behavioral: Trier Social Stress Test (TSST)
- Fludrocortisone & Placebo-TSST- BPD patients (Experimental): intake of 0.4mg fludrocortisone (orally) before "no stress"
  Interventions: Drug: Fludrocortisone; Behavioral: Placebo Trier Social Stress Test (P-TSST)
- Fludrocortisone & Placebo-TSST - Healthy controls (Experimental): intake of 0.4mg fludrocortisone (orally) before "no stress"
  Interventions: Drug: Fludrocortisone; Behavioral: Placebo Trier Social Stress Test (P-TSST)
- Placebo pills & Placebo-TSST - BPD patients (Experimental): intake of placebo pill before "no stress"
  Interventions: Behavioral: Placebo Trier Social Stress Test (P-TSST)
- Placebo pills & Placebo-TSST - Healthy controls (Experimental): intake of placebo pill before "no stress"
  Interventions: Drug: Placebo; Behavioral: Placebo Trier Social Stress Test (P-TSST)

INTERVENTIONS:
Drug: Fludrocortisone — pill of fludrocortisone
  Arms: Fludrocortisone & Placebo-TSST - Healthy controls; Fludrocortisone & Placebo-TSST- BPD patients; Fludrocortisone & TSST - BPD patients; Fludrocortisone & TSST - Healthy controls
Drug: Placebo — placebo pill
  Arms: Placebo pills & Placebo-TSST - Healthy controls; Placebo pills & TSST - BPD patients; Placebo pills & TSST - Healthy controls
Behavioral: Trier Social Stress Test (TSST) — psychosocial stress induction
  Other Names: Stress
  Arms: Fludrocortisone & TSST - BPD patients; Fludrocortisone & TSST - Healthy controls; Placebo pills & TSST - BPD patients; Placebo pills & TSST - Healthy controls
Behavioral: Placebo Trier Social Stress Test (P-TSST) — control condition
  Other Names: no stress
  Arms: Fludrocortisone & Placebo-TSST - Healthy controls; Fludrocortisone & Placebo-TSST- BPD patients; Placebo pills & Placebo-TSST - BPD patients; Placebo pills & Placebo-TSST - Healthy controls

SUMMARY:
The investigators will examine how a combination of pharmacological mineralocorticoid receptor (MR) stimulation and psychosocial stress will influence prosocial behavior in patients with Borderline Personality Disorder (BPD) compared to healthy controls (HC).

DETAILED DESCRIPTION:
The investigators will examine whether MR stimulation enhances prosocial behavior in BPD patients under additional psychosocial stress. Participants will be randomly assigned to receive either fludrocortisone as an MR stimulant or placebo. Afterwards, participants will either undergo the stress or placebo condition of the Trier Social Stress Test ((P-)TSST). Subsequently, cognitive and emotional empathy, as well as sharing and punishment behavior will be measured.

ELIGIBILITY:
Inclusion Criteria "BPD group":

* clinical diagnosis of borderline personality disorder
* female
* BMI between 17.5-30

Inclusion Criteria "control group":

* female
* BMI between 17.5-30
* no clinical diagnosis of any mental disorder

Exclusion Criteria:

* acute depressive episode,
* acute or lifetime psychotic symptoms
* acute substance abuse
* physical illness

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 240 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Empathy: Multifaceted Empathy Test | 15 minutes after (P-)TSST
  correct answers (mental state of the subject in the photos), rating of own emotional reaction

SECONDARY OUTCOMES:
Sharing behavior | 10 minutes after (P-)TSST
  amount of monetary units (max 100) shared with co-player
Punishment behavior | 10 minutes after (P-)TSST
  number of rejected offers from co-player

OTHER OUTCOMES:
salivary cortisol | 3 hours
  treatment check
salivary alpha amylase | 3 hours
  treatment check
sex hormones | 3 hours
  testosterone, estrogen, progesterone

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided